CLINICAL TRIAL: NCT02868099
Title: A Multi-center, Randomized, Placebo-controlled, Double-blinded Then Open 2 Stages Clinical Trial to Evaluate the Efficacy and Safety of Romiplostim in Adult Subjects With Persistent or Chronic Primary Immune Thrombocytopenia (ITP)
Brief Title: Efficacy and Safety of Romiplostim in Adult Subjects With Persistent or Chronic Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin China Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 531-CN002
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — romiplostim

STUDY DESIGN:
Intervention Model Description: multi-center, Randomized, Placebo-controlled, Double-blinded then Open-label
Who Masked: Participant, Investigator
Masking Description: Placebo-controlled, Double-blinded then Open-label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects received placebo for injection treatment will be administered subcutaneously once a week
  Interventions: Drug: Placebo
- Drug (Experimental): Subjects received Romiplostim for injection treatment will be administered subcutaneously once a week
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim
  Arms: Drug
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective is to evaluate the efficacy and safety of romiplostim for injection in adlut subjects with persistent or chronic primary immune thrombocytopenia (ITP).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with immune thrombocytopenia (ITP) for at least 6 months prior to signing the informed consent form (ICF).
* Subject is ≥ 18 years old while signing the ICF.
* Patients who have no response or relapsed after splenectomy. Or patients who have not been splenectomised and have no response or relapse to at least 1 prior treatment for immune thrombocytopenia (ITP).
* The mean of 3 scheduled platelet counts taken during the screening period must be: < 30 ×10^9/L, with none >35×10^9/L.

Exclusion Criteria:

* Any known history of bone marrow stem cell disorder. Any abnormal bone marrow findings other than those typical of ITP.
* Any active malignancy. If prior history of cancer other than basal cell carcinoma or cervical carcinoma in situ, and no treatment or active disease within 5 years prior to signing the ICF..
* Received hematopoietic growth factors (e.g., granulocyte colony-stimulating factor, macrophage colony-stimulating factor, erythropoietin, interleukin-11) for any reason within 4 weeks prior to signing the ICF.
* Received myeloproliferative leukemia (MPL) stimulation product other than the subject who had suspended recombinant human thrombopoietin (rHuTPO) for injection for 4 weeks before signing ICF.
* Received any anti-malignancy agents (e.g., cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, Interferon-alfa) for any reason within 8 weeks prior to signing the ICF.
* Received any monoclonal antibody drugs (e.g., rituximab) for any reason within 14 weeks prior to signing the ICF.
* Less than 4 weeks since end of any clinical trials about therapeutic drug or device prior to signing the ICF.
* Pregnant or breastfeeding.
* In the opinions of the principal investigator or investigators, the patients are not suitable for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of weeks in which the platelet response counts increase above 50×10^9/L | 6 weeks

SECONDARY OUTCOMES:
Proportion of subjects whose platelet counts relative to the baseline increase ≥ 20×10^9/L | 6 weeks
Proportion of subjects who have received emergency treatment to increase the platelet counts | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peking Union Medical College Hospital,, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou H, Zhou J, Wu D, Ma L, Du X, Niu T, Yang R, Liu J, Zhang F, Shi Q, Wang X, Jing H, Li J, Wang X, Cui Z, Zhou Z, Hou M, Shao Z, Jin J, Li W, Ren H, Hu J, Shen J, Liu L, Zeng Y, Zhou J, Liu X, Shen Y, Ding K, Taira T, Cai H, Zhao Y. Romiplostim in primary immune thrombocytopenia that is persistent or chronic: phase III multicenter, randomized, placebo-controlled clinical trial in China. Res Pract Thromb Haemost. 2023 May 23;7(5):100192. doi: 10.1016/j.rpth.2023.100192. eCollection 2023 Jul. PMID 37601010